CLINICAL TRIAL: NCT00356304
Title: Antidepressant Adherence Among Hispanics: A Motivational Interviewing Approach
Brief Title: Motivational Interviewing to Improve Medication Adherence Among Hispanic Adults With Depression
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Medicine and Dentistry of New Jersey (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Alejandro Interian, Ph.D., Adjunct Assistant Professor, National Institute of Mental Health (NIMH)
Organization: Rutgers, The State University of New Jersey (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: K23MH074860 (NIH); K23MH074860 (NIH); DSIR 8K-RT
Record Dates: First submitted 2006-07-21; First posted 2006-07-25 (Estimated); Results first posted 2014-05-08 (Estimated); Last update posted 2014-05-08 (Estimated); Status verified 2014-04

CONDITIONS: Depression
Keywords: Dysthymia; Major Depression; Hispanics; Latinos; Motivational Interviewing; Adherence
MeSH Terms: conditions — Depression; Dysthymic Disorder; Depressive Disorder, Major | interventions — Motivational Interviewing; Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Participants will receive motivational interviewing in addition to their antidepressant therapy
  Interventions: Behavioral: Motivational interviewing
- 2 (Active Comparator): Participants will receive treatment as usual
  Interventions: Behavioral: Treatment as usual

INTERVENTIONS:
Behavioral: Motivational interviewing — Participants assigned to motivational interviewing will attend two 1-hour sessions of motivational interviewing over 2 consecutive weeks, followed by a third session 8 weeks later. Motivational interviewing is a type of counselling. Each session is of approximately 1 hour duration.
  Arms: 1
Behavioral: Treatment as usual — Participants will continue with their normal treatment regimen as usual.
  Arms: 2

SUMMARY:
This study will determine the effectiveness of motivational interviewing in improving antidepressant medication adherence among Hispanics.

DETAILED DESCRIPTION:
Depression is a serious mental illness characterized by symptoms that can interfere with a person's ability to work, study, eat, sleep, and enjoy activities that were once pleasurable. Studies have shown that people of Hispanic descent tend to underutilize mental health care services. Additionally, Hispanics have demonstrated lower compliance and completion rates for antidepressant treatment. This may be due to low socioeconomic status, lack of family financial support, and inadequate communication with mental health care providers. Motivational interviewing is a goal-oriented type of therapy that focuses on eliciting behavior change by identifying and mobilizing a person's values. This study will determine the effectiveness of culturally sensitive motivational interviewing in improving antidepressant medication adherence in Hispanics.

Participants in this 6-month, open-label study will be randomly assigned to receive either motivational interviewing in addition to their antidepressant therapy or treatment as usual. All participants will first attend a 45-minute screening visit, which will include questionnaires and an interview about psychiatric symptoms, medication attitudes, and medication adherence behavior. Participants will also receive an electronic medication container that will record how consistently medication is taken. Participants assigned to motivational interviewing will then attend two 1-hour sessions of motivational interviewing over 2 consecutive weeks, followed by a third session 8 weeks later. The group assigned to treatment as usual will not partake in motivational interviewing, but will continue to receive their normal care. All participants will return to the study site for follow-up assessments, which will include measures of antidepressant adherence, at Months 2 and 5.

ELIGIBILITY:
Inclusion Criteria:

* Self-identifies as Hispanic
* DSM-IV diagnosis of any unipolar depressive disorder (i.e., MDD, dysthymia, or depressive disorder not otherwise specified)
* Currently taking antidepressant medication

Exclusion Criteria:

* Clinically significant suicidal ideation
* DSM-IV diagnosis of any substance-related disorder, bipolar disorder, or psychotic disorder/features within 12 months prior to study entry
* Unstable general medical condition

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2006-04; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alejandro Interian, PhD, Principal Investigator — Rutgers, The State University of New Jersey
Locations (1):
- University Behavioral Healthcare, New Brunswick, New Jersey, United States

REFERENCES:
- [Background] Interian A, Martinez IE, Guarnaccia PJ, Vega WA, Escobar JI. A qualitative analysis of the perception of stigma among Latinos receiving antidepressants. Psychiatr Serv. 2007 Dec;58(12):1591-4. doi: 10.1176/ps.2007.58.12.1591. PMID 18048562
- [Background] Escobar JI, Cook B, Chen CN, Gara MA, Alegria M, Interian A, Diaz E. Whether medically unexplained or not, three or more concurrent somatic symptoms predict psychopathology and service use in community populations. J Psychosom Res. 2010 Jul;69(1):1-8. doi: 10.1016/j.jpsychores.2010.01.001. Epub 2010 Feb 16. PMID 20630257
- [Result] Interian A, Lewis-Fernandez R, Gara MA, Escobar JI. A randomized-controlled trial of an intervention to improve antidepressant adherence among Latinos with depression. Depress Anxiety. 2013 Jul;30(7):688-96. doi: 10.1002/da.22052. Epub 2013 Jan 8. PMID 23300127

RESULTS

PARTICIPANT FLOW:
Groups:
- Motivational Enhancement Therapy for Antidepressants: Participants in this condition received TAU that was enhanced with three sessions of META. Two sessions were provided between the time 1 and time 2 evaluations, with a booster session occurring between the time 2 and time 3 evaluations. These participants were also receiving psychopharmacologic/psychotherapeutic care that was naturalistic.
- Treatment as Usual: Participants in this condition received usual care provided at the bilingual division of the CMHC. This included medication management, as well as some psychotherapy treatment. All aspects of care for participants in TAU was naturalistic and determined by CMHC psychiatrists and therapists who were not part of the study.
Period: Overall Study
Arm/Group | Motivational Enhancement Therapy for Antidepressants | Treatment as Usual
Started | 26 | 24
Completed | 24 | 20
Not Completed | 2 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Motivational Enhancement Therapy for Antidepressants | Treatment as Usual | Total
Number analyzed (Participants) | 26 | 24 | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.2 (10.8) | 41 (13) | 40.6 (11.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 19 | 38
  Male | 7 | 5 | 12
Region of Enrollment [Number; unit: participants]
  United States | 26 | 24 | 50

OUTCOME MEASURES:

1. Primary Outcome: Medication Adherence, as Measured by Electronic Pill Container
Description: Medication container caps (MEMS) recorded each instance where the antidepressant medication container was opened. An adherence index was derived the represented the percentage of days, within the medication period, where the container was opened.
Time Frame: Measured immediately post-treatment and at Months 2 and 5 months follow-ups
Population: We used an ITT with LOCF. These figures represent outcomes at 5 months.
Measure: Mean (Standard Error); unit: Percentage of Days
Arm/Group | Motivational Enhancement Therapy for Antidepressants | Treatment as Usual
Number analyzed (Participants) | 26 | 24
Percentage of Days | 58.76 (6.59) | 34.7 (6.87)
Statistical Analysis 1: Comparison: Motivational Enhancement Therapy for Antidepressants vs Treatment as Usual; Test type: Superiority or Other; p < .05, ANCOVA

2. Secondary Outcome: Treatment Retention
Time Frame: Measured at Month 5
Reporting Status: Not Posted

3. Secondary Outcome: Beck Depression Inventory-II (BDI-II)
Description: The BDI-II contains 21 questions, each answer being scored on a scale value of 0 to 3.
  0-13: minimal depression; 14-19: mild depression; 20-28: moderate depression; and 29-63: severe depression. Higher total scores indicate more severe depressive symptoms.
Time Frame: Measured at Month 5
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Motivational Enhancement Therapy for Antidepressants | Treatment as Usual
Number analyzed (Participants) | 26 | 24
units on a scale | 16.75 (2.70) | 23.03 (2.81)

4. Secondary Outcome: Medication Attitudes
Time Frame: Measured at Month 5
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Motivational Enhancement Therapy for Antidepressants | Treatment as Usual
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/24
Other Adverse Events (participants affected / at risk) | 0/26 | 0/24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No